CLINICAL TRIAL: NCT01905397
Title: Evaluation of Negative Pressure Wound Therapy for Reduction of Postoperative Surgical Site Infection in Patients Undergoing Colorectal and Hepatopancreatobiliary Surgery
Brief Title: Negative Pressure Wound Therapy to Reduce Surgical Site Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Kinetic Concepts, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00045975
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Results first posted 2022-10-10 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Patients Undergoing Hepatopancreatobiliary Surgery
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Negative Pressure Wound Therapy (Active Comparator): The Prevena Incision Management System is a 510K cleared device that covers and protects the incision from external infectious sources, while negative pressure removes fluid and infectious material from the surgical incision. The ActiVAC pump (also 510K cleared) may be used in some cases with the Prevena dressings as to achieve the negative pressure
  Interventions: Device: Negative pressure wound therapy
- Conventional wound therapy (Active Comparator): Traditional wound therapy (sterile bandages and dressing)
  Interventions: Device: Conventional wound therapy

INTERVENTIONS:
Device: Conventional wound therapy — Sterile bandages and wound coverings
  Arms: Conventional wound therapy
Device: Negative pressure wound therapy — The Prevena Incision Management System covers and protects the incision from external infectious sources, while negative pressure removes fluid and infectious material from the surgical incision. The ActiVAC pump may be used with the Prevena dressings as well in some situations to achieve negative pressure.
  Other Names: Prevena Incision Management System; ActiVAC
  Arms: Negative Pressure Wound Therapy

SUMMARY:
The purpose of this study is to compare the rate of surgical site infection between traditional wound care and negative pressure wound therapy. Wounds will be assessed 4-5 days after surgery and at the first clinic visit after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients 18 years of age or older
* Scheduled for an elective surgery in either open CRS or open HPBS. This includes, but is not limited to: ileocecectomy, right hemicolectomy, extended right hemicolectomy, transverse colectomy, left hemicolectomy, sigmoidectomy, proctectomy, low anterior resection, or abdominoperineal resection gastrectomy, hepatectomy, bile duct reconstruction, duodenectomy, pancreatectomy, pancreaticoduodenectomy, or pancreatic duct reconstruction

Exclusion Criteria:

* The need for emergency surgery.
* The need for use of only laparoscopic surgery.
* Presence of bowel obstruction, strangulation, peritonitis or perforation.
* The presence of local or systemic infection preoperatively.
* ASA class ≥4.
* Inability to provide informed consent and authorization.
* Known allergy or hypersensitivity to silver.
* Any clinically significant condition that, in the investigator's opinion, would significantly impair the subject's ability to comply with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2013-12-18 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Blazer, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ceppa EP, Kim RC, Niedzwiecki D, Lowe ME, Warren DA, House MG, Nakeeb A, Zani S, Moyer AN, Blazer DG 3rd; Closed Incision Negative Pressure Therapy (ciNPT) Investigators. Closed Incision Negative Pressure Therapy to Reduce Surgical Site Infection in High-Risk Gastrointestinal Surgery: A Randomized Controlled Trial. J Am Coll Surg. 2023 Apr 1;236(4):698-708. doi: 10.1097/XCS.0000000000000547. Epub 2023 Jan 10. PMID 36728375

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at Duke University Medical Center from December 18, 2013 to April 8, 2021 and at Indiana University from December 12, 2016 to April 8, 2021.
Groups:
- Conventional Wound Therapy: Sterile bandages and dressings.
Period: Overall Study
Arm/Group | Negative Pressure Wound Therapy | Conventional Wound Therapy
Started | 82 | 82
Completed | 63 | 75
Not Completed | 19 | 7
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Surgery canceled/aborted | 9 | 5
Not completed — Incision < 7 cm | 2 | 0
Not completed — Wrong treatment | 1 | 1
Not completed — Device not applied | 3 | 0
Not completed — Dressing not applied in operating room | 1 | 0
Not completed — Wound vac turned off due to device alarm | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Negative Pressure Wound Therapy | Conventional Wound Therapy | Total
Number analyzed (Participants) | 82 | 82 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (10.1) | 61.1 (12.3) | 61.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 44 | 91
  Male | 35 | 38 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 76 | 78 | 154
  Unknown or Not Reported | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 8 | 21
  White | 65 | 69 | 134
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Participants With a Surgical Site Infection
Description: Number and percentage of participants with at least 1 surgical site infection (SSI).
Time Frame: 30 days after surgery; assessed at 4-5 days and 30 days post-operation
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Negative Pressure Wound Therapy | Conventional Wound Therapy
Number analyzed (Participants) | 63 | 75
Participants | 14 | 20
Statistical Analysis 1: Comparison: Negative Pressure Wound Therapy vs Conventional Wound Therapy; Test type: Superiority; p = 0.27, t-test, 1 sided; Difference in proportions = 0.05

2. Secondary Outcome: Number of Surgical Site Infections by Type
Description: Each surgical site infection was classified into one of the following categories: superficial incisional, deep incisional, or organ/space (as defined by The American College of Surgeons NSQIP [National Surgical Quality Improvement Program] guidelines). The number of infections in each category is reported separately for both treatment arms. Some participants had multiple infections.
Time Frame: 30 days post-surgery
Measure: Count of Units; unit: infections
Units Other Than Participants: infections
Arm/Group | Negative Pressure Wound Therapy | Conventional Wound Therapy
Number analyzed (Participants) | 63 | 75
Number analyzed (infections) | 16 | 23
infections
  Superficial Incisional | 7 | 7
  Deep Incisional | 2 | 6
  Organ/Space | 7 | 10

3. Secondary Outcome: Length of Hospital Stay
Description: Assess (or compare) the length of hospital stay between subjects who receive standard of care and incisional V.A.C. via PIMS.
Time Frame: Up to 62 days post-surgery
Measure: Median (Full Range); unit: days
Arm/Group | Negative Pressure Wound Therapy | Conventional Wound Therapy
Number analyzed (Participants) | 63 | 75
days | 8 [3 to 46] | 6 [3 to 62]

ADVERSE EVENTS:
Time Frame: 30 days after surgery
Arm/Group | Negative Pressure Wound Therapy | Conventional Wound Therapy
All-Cause Mortality (participants affected / at risk) | 0/63 | 1/75
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/75
Other Adverse Events (participants affected / at risk) | 1/63 | 0/75
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Negative Pressure Wound Therapy (N=63) | Conventional Wound Therapy (N=75)
Rash, Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-31): https://cdn.clinicaltrials.gov/large-docs/97/NCT01905397/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/97/NCT01905397/ICF_001.pdf